CLINICAL TRIAL: NCT03292861
Title: A Pilot Randomized Study to Assess the Effect and Safety Profile of Thymoglobulin® in Primary Cardiac Transplant Recipients: A 12-month, Single Center, Randomized, Open-label Study of Efficacy Comparing Immediate Treatment With and Without Thymoglobulin® 1.5 mg/kg/d for 5 Consecutive Days in Heart Transplant Recipients
Brief Title: The Effect and Safety Profile of Thymoglobulin® in Primary Cardiac Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Principal Investigator, Jon Kobashigawa, Director of Advanced Heart Disease Program, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ATG Pilot Study
Record Dates: First submitted 2017-09-12; First posted 2017-09-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — thymoglobulin; Mycophenolic Acid; Tacrolimus; Sirolimus; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Thymoglobulin® (Active Comparator): Thymoglobulin® (Genzyme) [rabbit anti-thymocyte globulin (ATG)] is a purified pasteurized, gamma immune globulin, obtained by immunization of rabbits with human thymocytes. This immunosuppressive product contains polyclonal cytotoxic antibodies directed against antigens expressed on human T-lymphocytes. Approximately half of the patients will be randomized to receive a total of 5 doses of Thymoglobulin during the study. The first dose of Thymoglobulin will be administered at 1.5 mg/kg via intravenous infusion over 6 hours immediately upon arrival to the ICU post-operation (day 1). Subsequent doses of 1.5 mg/kg will be administered on days 2, 3, 4, and 5 via IV infusion over 4 hours.
  In addition, there will be maintenance doses of mycophenolate mofetil, tacrolimus, sirolimus, and cumulative dose of corticosteroids at 12 months post-transplantation
  Interventions: Drug: Thymoglobulin; Drug: Mycophenolate Mofetil; Drug: Tacrolimus; Drug: Sirolimus; Drug: Corticosteroids
- No induction therapy (No Intervention): Patients qualifying for the study will be randomized before the transplantation surgery in a 1:1 ratio to either Thymoglobulin® or no treatment.

INTERVENTIONS:
Drug: Thymoglobulin — Approximately half of the patients will be randomized to receive a total of 5 doses of Thymoglobulin during the study. The first dose of Thymoglobulin will be administered at 1.5 mg/kg via intravenous infusion over 8 hours immediately upon arrival to the ICU post-operation (day 1). Subsequent doses of 1.5 mg/kg will be administered on days 2, 3, 4, and 5 via IV infusion over 4-8 hours.
  Arms: Thymoglobulin®
Drug: Mycophenolate Mofetil — 3.0 grams divided bid begun post-transplant, either IV or po as tolerated by patient. Initial dose must be given within 24 hours post-transplant. Dosing will be titrated based on recipient's body size and any adverse side effects
  Arms: Thymoglobulin®
Drug: Tacrolimus — Doses of 1-4 mg bid either IV or po will be prescribed to achieve a target trough level of 10-15 ng/mL before post-operative day number 5. Target trough levels are 10-15 ng/mL for post-operative days #1-30, 8-12ng/mL days#31-60 and 5-10 ng/mL thereafter.
  Arms: Thymoglobulin®
Drug: Sirolimus — Maintenance doses of sirolimus at 12 months post-transplantation
  Arms: Thymoglobulin®
Drug: Corticosteroids — 125 mg IV methylprednisolone immediately post-operatively x 3 doses q12hrs, then switching to oral prednisone at 1.0 mg/kg/day po divided into bid doses that are rounded off to the next higher 5 mg increment. For example, a 76 kg person would should be dosed at 38 mg po bid, which rounded off to the next 5 mg increment would be 40 mg po bid. (Equivalent dosing via an alternative route may be used if pos not tolerated or contraindicated). Prednisone will be tapered by 10 mg qd until the dose of 10 mg po bid is reached.
  Arms: Thymoglobulin®

SUMMARY:
This is a randomized, controlled, single center study to evaluate the efficacy of Thymoglobulin induction therapy in combination with Mycophenolate Mofetil, tacrolimus, and steroids in the prevention of CAV. Approximately half of the patients will be randomized to receive a total of 5 doses of Thymoglobulin during the study. The first dose of Thymoglobulin will be administered at 1.5 mg/kg via intravenous infusion over 6 hours immediately upon arrival to the ICU post-operation (day 1). Subsequent doses of 1.5 mg/kg will be administered on days 2, 3, 4, and 5 via IV infusion over 4 hours.

Mechanistic assays (T-reg cells, Lym subsets, B cell subsets, IL-1b, cytokines, TGFb, IL-21 to be drawn at Pre-transplant, 3, 6, 12 months post-transplant) will also be performed.

All patients will be followed and monitored according to standard of care protocols for heart transplant recipients at our center.

ELIGIBILITY:
Inclusion Criteria for Study Entry:

1. Subjects must be undergoing their first allograft transplant
2. Men and non-pregnant women must be 18 to 70 years old
3. Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to transplantation. The sensitivity must be equal to at least 50 mIU/mL. (Urine test is allowed in addition to serum test in patients where serum results are delayed)
4. Men with a female partner of child bearing age and women of childbearing potential must use two reliable forms of contraception simultaneously. Effective contraception must be used before beginning study drug therapy, and for 4 months following discontinuation of study drug therapy.
5. Subjects must be willing and capable of understanding the purpose and risks of the study, and must sign a statement of informed consent
6. Subjects with a Creatinine < 2.0 mg/dl at time of transplant

Exclusion Criteria for Study Entry:

1. Allergy to Thymoglobulin-Thymoglobulin is contraindicated in patients with history of allergy or anaphylaxis to rabbit proteins or to any product excipients, or who have active acute or chronic infections which contraindicate any additional immunosuppression
2. Previous organ transplants
3. Patients receiving multiple organs
4. Patients with a BMI higher than 35
5. Patients with PRA ≥ 25%
6. Patients requiring VAD upon completion of transplantation surgery.
7. HIV-1, HTLV-1, chronic Hepatitis B, or chronic Hepatitis C infection
8. Documented or strong suspicion for pre-operative active infection that has not yet been adequately treated with the recommended course of antimicrobial therapy
9. Presence of any chronic myelosuppressive disease or agent that has resulted in either chronic leucopenia or chronic thrombocytopenia
10. Active peptic ulcer disease and active GI bleeding
11. Patients who have received within the past 30 days or require concomitant treatment with other investigational drugs (except for those listed in section 8.6 "Concomitant treatment")
12. Patients with a history of AL amyloidosis (TTR amyloids) are permitted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Composite Efficacy Failure at 12 Months | 12 Months
  Composite efficacy failure is defined as development of de novo donor specific antibodies (measured by standardized alloantibody testing by Luminex and control sera, characterizing kinetics, specificities and relative binding strength) and ischemia on endomyocardial biopsy (characterized on biopsy by myocyte necrosis and/or regions of myocyte dropout) at 12 months post-transplant.

SECONDARY OUTCOMES:
Changes in immune cell profiles | 12 months
  Correlations between significant changes in immune cell profiles and biomarkers, and their relation to any significant differences in clinical outcomes
Changes in biomarkers | 12 months
  Correlations between significant changes in biomarkers and their relation to any significant differences in clinical outcomes
Number of patients who experience rejection | 12 months
  Number of patients who experience acute cellular, antibody-mediated, hemodynamic compromise, and any-treated rejection within first 12 months after transplantation/
Number of episodes per patient | 12 months
  Number of acute cellular, antibody-mediated, hemodynamic compromise and any-treated rejection episodes per patient within the first 12 months post-transplantation
First rejection by ISHLT biopsy grading scale | 12 months
  First acute cellular, antibody-mediated, hemodynamic compromise, and any-treated rejection by the ISHLT biopsy grading scale in the first 12 months post-transplantation
Time to first rejection | 12 months
  Time to first acute cellular, antibody-mediated, hemodynamic compromise, and any-treated rejection within the first 12 months
Incidence of primary graft dysfunction (PGD) | first 24 hours post-transplant
  The incidence of Primary Graft Dysfunction(PGD) in the first 24 hours post-transplant
Patient and graft survival | 12 months
  Patient and graft survival at 12 months post-transplantation
Types of patients with fatal infectious complications | 12 months
  The types of patients with fatal infectious complications (especially CMV infection) within the first 12 months post-transplantation
Number of patients with fatal infectious complications | 12 months
  The number of patients with fatal infectious complications (especially CMV infection) within the first 12 months post-transplantation
Types of patients with non-fatal infectious complications | 12 months
  Types of patients with non-fatal infectious complications (especially CMV infection) within the first 12 months post-transplantation
Number of patients with non-fatal infectious complications | 12 months
  Number of patients with non-fatal infectious complications (especially CMV infection) within the first 12 months post-transplantation
Freedom from development of circulating antibodies | 12 months
  Freedom from the development of circulating antibodies within the first 12 months post transplantation, where circulating antibodies include donor specific antibodies (DSA), non-specific antibodies, and non-human leukocyte antigen antibodies
Change in coronary maximal intimal thickness | 12 months
  Change in coronary maximal intimal thickness at matched sites by intravascular ultrasound at 12 months
Change in coronary intimal area | 12 months
  Change in coronary intimal area at matched sites by intravascular ultrasound at 12 months
Change in coronary intimal volume | 12 months
  Change in coronary intimal volume at matched sites by intravascular ultrasound at 12 months
Change in coronary vessel area | 12 months
  Change in coronary vessel area at matched sites by intravascular ultrasound at 12 months
Change in coronary intimal index | 12 months
  Change in coronary intimal index at matched sites by intravascular ultrasound at 12 months
Change in coronary percent atheroma volume | 12 months
  Change in coronary percent atheroma volume at matched sites by intravascular ultrasound at 12 months
Maintenance doses of mycophenolate mofetil, tacrolimus, sirolimus, and dose of corticosteroids | 12 months
  Maintenance doses of mycophenolate mofetil, tacrolimus, sirolimus, and cumulative dose of corticosteroids at 12 months post-transplantation
Number of hospital days per patient | 3 months, 6 months, 12 months
  Number of hospital days per patient, both during the transplant period and during the post-transplant period at 3 months, 6 months, and 1 year
Number of patients requiring hospitalization | 3 months, 6 months, 12 months
  Number of patients requiring hospitalization by 3 months, by 6 months, or by 1 year post-transplantation
Death/Re-transplant | 12 months
  To describe between treatment groups the incidence of the composite primary endpoint of death/re-transplant at 12 months post-transplantation
Hemodynamic compromise rejection | 12 months
  To describe between treatment groups the incidence of the composite primary endpoint of hemodynamic compromise rejection at 12 months post-transplantation. This is an ejection fraction of ≤ 30% or a 0.20 absolute decrease from baseline, and the need for inotropic agents OR a fractional shortening ≤ 20% or a 25% decrease from baseline, and the need for inotropic agents PLUS need for inotropic agents due to a Cardiac Index (CI) < 2.0 L/min/m2 or a 25% decrease from baseline
Graft dysfunction | 12 months
  To describe between treatment groups the incidence of the composite primary endpoint of graft dysfunction (ejection fraction less than or equal to 40% by echocardiography)at 12 months post-transplantation
Cellular rejection | 12 months
  To describe between treatment groups the incidence of the composite primary endpoint of biopsy proven cellular rejection ≥2R at 12 months post-transplantation
Antibody mediated rejected | 12 months
  To describe between treatment groups the incidence of the composite primary endpoint of biopsy proven antibody mediated rejection ≥AMR1 at 12 months post-transplantation
Cardiac Allograft Vasculopathy (CAV) | 12 months
  To describe between treatment groups the incidence of cardiac allograft vasculopathy (CAV) (defined as a change ≥0.5mm in maximal intimal thickness (MIT) of the coronary arteries by intravascular ultrasound at 12 months as compared to baseline)
Any treated rejection | 12 months
  To describe between treatment groups any treated rejection at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon Kobashigawa, MD, Principal Investigator — Director
Locations (2):
- United States (2):
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California

DOCUMENTS (1):
  • Study Protocol (2023-08-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT03292861/Prot_001.pdf